CLINICAL TRIAL: NCT03906500
Title: High Schools- High on Life: an Intervention to Reduce Excessive Drinking in Danish High Schools
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the corona-crisis, we asses that it is not possible to carry out the effect-measurement as planned. The lockdown has strongly affected the young people's social life and alcohol use that could hide possible effects of the intervention.
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Veronica Pisinger, Research assistent, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15/4155_2
Record Dates: First submitted 2019-03-29; First posted 2019-04-08 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Drinking
Keywords: Adolescence; Alcohol use; High school
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: The study will employ a cluster-randomized controlled study design: investigators plan to include a random sample of at least 12 high schools randomly 1:1 allocated to either intervention or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consist of three main components.
  School environmental component
  The component targeting the high school environment consisted of two separate elements:
  * Revision of school alcohol policy
  * Appointment of coordinator(s) of student committees organizing events, where alcohol is sold, and student introduction committee.
  Student components
  The Student components consisted of three main elements:
  * Web-based education for the student committees organizing events where alcohol is sold and the student introduction committee
  * Pocket movie campaign
  * Social norms campaign
  Parent components
  The parent component consisted of three separate elements:
  * Parent Information Meeting
  * Parent Information Folder
  * Parent Information Website
  Interventions: Behavioral: High schools High on Life
- control group (No Intervention): Control high schools was asked to continue business as usual and promised to receive the intervention in the school year starting in 2020

INTERVENTIONS:
Behavioral: High schools High on Life — The intervention consist of three main components.
  Environmental factors of the school environment
  The component targeting the high school environment consisted of two separate elements:
  * Revision of school alcohol policy
  * Appointment of coordinator(s) of student committees organizing events, where alcohol is sold, and student introduction committee.
  Student component
  The Student components consisted of three main elements:
  * Online education for the student committees organizing events where alcohol is sold and the student introduction committee
  * Pocket movie campaign competition
  * Social norms campaign
  Parent component
  The parent component consisted of three separate elements:
  * Parent Information Meeting
  * Parent Information Folder
  * Parent Information Website
  Arms: Intervention

SUMMARY:
High schools High on life' intervention is a high school-based, multi-component intervention guided by theory, evidence, and empirical findings to reduce excessive drinking among Danish high school students. The study will employ a cluster-randomized controlled study design: investigators plan to include a random sample of at least 12 high schools randomly 1:1 allocated to either intervention or control group. Timeline: Baseline data will be obtained from the Danish National Youth Study 2019, collected in January to March 2019. Delivery of intervention: August 2019 to January 2020. Follow-up survey: April to May 2020. Primary outcome measure: mean number of binge-drinking episodes within the last 30 days. Secondary outcome measures: weekly alcohol consumption, alcohol intake at last school party, alcohol intake at the school during last school party, number of students that agrees that they are able to have fun at a party without drinking, and the proportion of students that think alcohol plays a too dominant part at the school. Implementation will be monitored thorough process evaluation.

DETAILED DESCRIPTION:
High schools High on life' intervention is a high school-based, multi-component intervention guided by theory, evidence, and empirical findings to reduce excessive drinking among Danish high school students. The study will employ a cluster-randomized controlled study design: based on sample size calculations investigators plan to include a random sample of at least 12 high schools randomly 1:1 allocated to either intervention or control group.

Timeline: Baseline data will be obtained from the Danish National Youth Study 2019, collected in January to March 2019. Delivery of intervention: August 2019 to January 2020. Follow-up survey: April to May 2020. Primary outcome measure: mean number of binge-drinking episodes within the last 30 days. Secondary outcome measures: weekly alcohol consumption, alcohol intake at last school party, alcohol intake at the school during last school party, number of students that agrees that they are able to have fun at a party without drinking, and the proportion of students that think alcohol plays a too dominant part at the school. Implementation will be monitored thorough process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in High school that participate in The Danish National Youth Study 2019
* General High Schools

Exclusion Criteria:

* non General High schools students
* non participation in The Danish National Youth Study 2019

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3682 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Mean number of binge drinking occasions within the last 30 days | 12 months
  30% lower number of binge drinking occasions within the last 30 days

SECONDARY OUTCOMES:
Weekly alcohol consumption | 12 months
  Mean weekly alcohol consumption
Alcohol intake at last school party | 12 months
  Alcohol intake at last school party
Alcohol intake at the school during last school party | 12 months
  Alcohol intake at the school during last school party
Proportion that think alcohol play a too dominant part at the school | 12 months
  Proportion who think alcohol play a too dominant part at the school

OTHER OUTCOMES:
Social inclusion | 12 months
  Proportion of students who feel included in the social community at school, including students that do not drink or have a low alcohol intake
Marihuana use | 12 months
  proportion of students who have smoked marihuana
Other drug use | 12 months
  Proportion who have tried other drugs than marihuana

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Pisinger, Principal Investigator — the national institute of public health, Southern Denmark University
Locations (1):
- National Institute of Public Health, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pisinger VSC, Hoffmann SH, Palsson L, Dalum P, Gronbaek MK, Tolstrup JS, Thygesen LC, Krolner RF. 'High schools High on life': Development of an Intervention to Reduce Excessive Drinking in Danish High Schools. Front Public Health. 2020 Sep 15;8:435. doi: 10.3389/fpubh.2020.00435. eCollection 2020. PMID 33042935
- [Derived] Pisinger VSC, Hoffmann S, Rosing JA, Gronbaek M, Tolstrup JS, Thygesen L, Krolner R. Study protocol for a cluster randomised controlled trial testing the effectiveness of the 'High schools High on life' intervention on reducing excessive drinking in Danish high schools. BMJ Open. 2020 Aug 6;10(8):e038857. doi: 10.1136/bmjopen-2020-038857. PMID 32764089

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT03906500/Prot_SAP_001.pdf